CLINICAL TRIAL: NCT03551392
Title: Pilot Intervention With Near Infrared Stimulation: Revitalizing Cognition in Older Adults and Those With Parkinson Disease
Brief Title: Pilot Intervention With Near Infrared Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: McKnight Brain Research Foundation (Unknown); University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB201801152; OCR18061 (Other: University of Florida); PRO00020250 (Other: UFIRST)
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Aging
Keywords: Cognitive Aging; Photobiomodulation; Low Level Light Therapy; Near Infrared (NIR) Light; Neuromodulation
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: This is a blinded parallel group sham controlled pilot trial, with half the participants in each group randomized to the real NIR treatment and half to the sham treatment condition.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Research assistants who administer pre and post measures will be masked, as well as participants who receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NIR -Older Adult (Active Comparator): Older adult participants receive the Medx Console System and the Vielight 810 intranasal stand alone unit. These interventions occur during 16 lab sessions (1.5 hours each) during an 12 week period, plus daily 25 minute 'at home' intranasal stimulation interventions, 4 days each week.
  Interventions: Device: Medx Console System; Device: Vielight 810 intranasal stand alone unit
- No Dose NIR-Older Adult (Sham Comparator): Older adult participants receive the sham Medx Console System and the sham Vielight 810 intranasal stand alone unit, since the devices deliver no near infrared light. These sham interventions occur during 16 lab sessions (1.5 hours each) during an 12 week period, plus daily 25 minute 'at home' intranasal stimulation interventions, 4 days each week.
  Interventions: Device: Sham Medx Console System; Device: Sham Vielight 810 intranasal stand alone unit

INTERVENTIONS:
Device: Medx Console System — This intervention delivers near infrared (NIR) light using light emitting diodes applied to the head and via an intranasal applicator for a period of approximately 1.5 hours. A total of 16 sessions take place in the lab over 12 weeks.
  Other Names: Low Level Light Therapy; Photobiomodulation; Transcranial Near Infrared Stimulation
  Arms: NIR -Older Adult
Device: Sham Medx Console System — This intervention uses sham application of near infrared light (NIR) using light emitting diodes applied to the head and via an intranasal applicator for a period of approximately 1.5 hours. A total of 16 sessions take place in the lab over 12 weeks.
  Arms: No Dose NIR-Older Adult
Device: Vielight 810 intranasal stand alone unit — Daily at home intranasal NIR stimulation sessions, 25 minutes in duration, 4 days each week.
  Arms: NIR -Older Adult
Device: Sham Vielight 810 intranasal stand alone unit — Daily at home intranasal "sham" NIR stimulation sessions, 25 minutes in duration, 4 days each week.
  Arms: No Dose NIR-Older Adult

SUMMARY:
The current study will test whether age-related cognitive and mood changes in older adults and those will be affected by near infrared (NIR) stimulation. The overall hypothesis, drawn from previous literature, is that exposure to NIR stimulation will have positive effects on brain health and will result in better cognitive and mood performance.

DETAILED DESCRIPTION:
This is a multi-site pilot study of the efficacy of NIR stimulation for enhancing cognition and mood in nondemented older adults. Sites include the University of Florida and University of Arizona. Prior research suggests that NIR exposure may be neuroprotective and increases energy available to neurons. The current study will test whether age-related cognitive and mood changes in older adults will be affected by near infrared (NIR) stimulation.

The study team will randomize older adults into treatment groups and evaluate neuroimaging and cognitive outcome measures, before and after a 12-week intervention involving transcranial and intranasal NIR. The protocol will involve both " lab" and " home-based" NIR stimulation. The overall hypothesis, drawn from previous literature, is that exposure to NIR stimulation will have positive effects on brain health and will result in better cognitive and mood performance.

ELIGIBILITY:
Inclusion Criteria:

* No evidence of dementia or Mild Cognitive Impairment based on cognitive screening (i.e., Montreal Cognitive Assessment (MoCA) scores within normal limits for age , education, and sex using the NACC Uniform Data Set (UDS) norms or Dementia Rating Scale (DRS-2) scores <5thile), and age-appropriate delayed Story recall (i.e., WMS-III Logical Memory) and confrontation naming (Boston Naming Test)
* Able to provide informed consent and perform cognitive and mood measures on a computer
* At least 8th grade education and/or ability to read at 8th grade level
* Willingness to be randomized to Sham or Real intervention
* Can devote 12 weeks to the intervention, and additional time for pre and post testing
* On stable doses of major medications; Since some older adults with subjective memory complaints may be prescribed acetylcholinererase inhibitors or related medications by their primary care physicians (i.e., donepezil, rivastigmine, galantaominhe, memantime, or other potential memory-enhancing agent(s), we will not exclude them as long as they have been on stable medications for at least two months and plan to continue this medication during study participation.
* Normal functional behavior in terms of daily activities

Exclusion Criteria:

* Previous major strokes or other known significant brain abnormalities or diseases affecting cognition (i.e., multiple sclerosis, seizure disorder, brain surgery, moderate TBI, etc.). No history of brain surgery. Exceptions are a diagnosis of Parkinson's disease for the PD subgroup.
* Unstable and uncontrolled medical conditions (metabolic encephalopathy, HIV, moderate to severe kidney or liver disease)
* Current or past history of major psychiatric disturbance including schizophrenia, or active psychosis, bipolar disorder, current major depressive episode, current alcohol or substance abuse or history thereof within the past six months. The study team is not excluding individuals who are taking antidepressants or anti-anxiety medications, however, use of antidepressants and anxiolytics will be recorded and data will be analyzed in post-hoc analyses
* Use of antipsychotics, sedatives, or other medications with significant anticholinergic properties (due to potential influence on memory)
* Use of photo-sensitive medications such as steroids or retin-A within 15 days of the study intervention
* Diagnosis of active cancer
* Significant motor or visual disturbance that would prevent one from using a computer or detecting colors
* Previous participation in a cognitive training study within the last 3 months or current involvement in another study involving cognitive training or intervention at the time of participation
* Inability to undergo brain imaging due to claustrophobia or implants such as pacemakers, heart valves, brain aneurysm clips, orthodontics, non-removable body jewelry, or shrapnel containing ferromagnetic metal

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
ARENA, learning and memory change from baseline to post-testing | Baseline to one-week post intervention (approx Week 14)
  Spatial navigation and memory task yields a score consisting of percent time spent in the target quadrant during the probe trial.

SECONDARY OUTCOMES:
NIH Examiner, Verbal Fluency Domain Score change from baseline | Change in baseline to one-week post intervention (approx Week 14)
  The Verbal Fluency domain from the NIH Examiner involves speeded production of letter and semantic cued words. Verbal fluency composite score can range from -3.0 to 3.0, with higher scores corresponding to better fluency performance and negative scores indicating impairment. A change score will be calculated by subtracting the baseline scores from the post test scores.
NIH Examiner, Working Memory Domain score change from baseline | Change in baseline to one-week post intervention (approx Week 14)
  Computer based battery of working memory tasks that yields a composite score based on Dot Counting total score and d-prime measures from the N-back task. Composite score ranges from -3.0 to 3.0, with higher scores corresponding to better working memory performance. A change score will be calculated by subtracting the baseline scores from the post test scores.
NIH Examiner, Cognitive Control Domain score change from baseline to post-testing | Change in baseline to one-week post intervention (approx Week 14)
  The Cognitive Control domain from the NIH Examiner yields a composite score based on individual scores from the Flanker task, the Continuous Performance task, and the Set-Shifting task. Composite score ranges from -3.0 to 3.0, with higher scores corresponding to better cognitive control performance. A change score will be calculated by subtracting the baseline scores from the post test scores.
NIH Toolbox Emotion Negative Affect Scale change from baseline to post-testing | Baseline to one-week post-intervention (approx Week 14)
  The Negative Affect Scale from the NIH Toolbox Emotion module results in T-scores (mean=50, SD=10) for categories such as anger, sadness, and apathy. Scores below 40 indicate low levels of negative affect. Change scores will be calculated by subtracting the baseline scores from the post-test scores.
NIH Toolbox Emotion-Psychological Well Being Scale change from baseline | Change in baseline to one-week post intervention (approx Week 14)
  The Psychological Well-being Scale from the NIH Toolbox Emotion module results in T-scores (mean=50, SD=10) for categories such general life satisfaction, meaning and purpose, and positive affect. Scores below 40 indicate low levels of positive affect. Change scores will be calculated by subtracting the baseline scores from the post-test scores.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Bowers, Ph.D., Principal Investigator — University of Florida; Adam Woods, Ph.D., Principal Investigator — University of Florida; Gene Alexander, Ph.D., Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No